CLINICAL TRIAL: NCT03397615
Title: Effect of Vaginal Douching With Betadine Versus Non Douching Before CS for Prevention of Post Operative Infections
Brief Title: Effect of Vaginal Douching With Betadine Before CS for Prevention of Post Operative Infections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 16
Record Dates: First submitted 2018-01-06; First posted 2018-01-12 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Puerperal Infection
MeSH Terms: conditions — Puerperal Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Betadine douches (Active Comparator): subjects received a vaginal preparation with povidone-iodine solution immediately prior to caesarean delivery
  Interventions: Behavioral: Betadine douches
- Non betadine douches (No Intervention): subjects didnot received a vaginal preparation prior to caesarean delivery

INTERVENTIONS:
Behavioral: Betadine douches — subjects received a vaginal preparation with povidone-iodine solution immediately prior to caesarean delivery
  Arms: Betadine douches

SUMMARY:
The present study was a prospective randomized controlled trial in which subjects received a vaginal preparation with povidone-iodine solution immediately prior to caesarean delivery or received no vaginal preparation

DETAILED DESCRIPTION:
The present study was a prospective randomized controlled trial in which subjects received a vaginal preparation with povidone-iodine solution immediately prior to caesarean delivery or received no vaginal preparation

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing CS

Exclusion Criteria:

* • Betadine allegy.

  * Rupture membranes.
  * Accidental Hemorrhage.
  * H/O suggestive chorioamnionitis ; uterine tenderness, offensive vaginal discharge, fever medical disorders as diabetes, hypertension , cardiac or renal diseqases

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 1200 (Estimated)
Dates: Start 2019-01-03 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Postpartum endometritis | 6 weeks after Cesarean section
  a clinical diagnosis, usually involving fever, uterine fundal tenderness, or prurulent lochia requiring antibiotic therapy.

SECONDARY OUTCOMES:
Postoperative wound infection | 6 weeks after Cesarean section
  erythema, tenderness, prurulent drainage from the incision site, with or without fever, requiring antibiotic therapy
Postoperative fever | 3 weeks after Cesarean section
  temperature higher than 38 degrees C

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Haas DM, Morgan S, Contreras K, Kimball S. Vaginal preparation with antiseptic solution before cesarean section for preventing postoperative infections. Cochrane Database Syst Rev. 2020 Apr 26;4(4):CD007892. doi: 10.1002/14651858.CD007892.pub7. PMID 32335895